CLINICAL TRIAL: NCT02525055
Title: A Randomised, Double Blind Study To Characterise Influenza A/Perth/16/2009(H3N2) Virus
Brief Title: Characterisation of a New Wild-Type H3N2 Virus for the Human Viral Challenge Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvivo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RVL-vCS-003
Record Dates: First submitted 2015-08-06; First posted 2015-08-17 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Influenza
Keywords: Flu; Influenza; Human Viral Challenge Model; Wild-Type; H3N2; Universal Influenza Vaccine; Intra-seasonal vaccines; Antiviral
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Cohort 1 (including 4 arms) is double blinded. Cohort 2 (including 1 arm divided in 2 separate age comparison groups) is open labelled. In order to allow for an age comparison between subjects aged 18 to 45 and subjects aged 56 to 64, data from Cohort 2 (Infectious Titre 5) will be presented in 2 separate reporting groups.
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Infectious titre 1 (Experimental): 6 participants aged 18 to 45 were inoculated with 1mL containing 2.8 x 10*3 TCID50 of virus
  Interventions: Other: Infectious titre 1 (H3N2)
- Infectious titre 2 (Experimental): 6 participants aged 18 to 45 were inoculated with 1mL containing 2.5 x 10*4 TCID50 of virus
  Interventions: Other: Infectious titre 2 (H3N2)
- Infectious titre 3 (Experimental): 6 participants aged 18 to 45 were inoculated with 1mL containing 3.6 x 10*5 TCID50 of virus
  Interventions: Other: Infectious titre 3 (H3N2)
- Infectious titre 4 (Experimental): 6 participants aged 18 to 45 were inoculated with 1mL containing 4.7 x 10*6 TCID50 of virus
  Interventions: Other: Infectious titre 4 (H3N2)
- Infectious titre 5 (age 18 to 45 y) (Experimental): 6 participants aged 18 to 45 were inoculated with 1mL containing 3.5 x 10*5 TCID50 of virus.
  Interventions: Other: Infectious titre 5 (H3N2) (Subjects aged 18 to 45 years old)
- Infectious titre 5 (age 46 to 64 y) (Experimental): 16 participants aged 46 to 64 were inoculated with 1mL containing 3.5 x 10*5 TCID50 of virus.
  Interventions: Other: Infectious titre 5 (H3N2) (Subjects aged 46 to 64 years old)

INTERVENTIONS:
Other: Infectious titre 1 (H3N2) — Infectious titre 1: 2.8 x 10*3 TCID50/mL
  Arms: Infectious titre 1
Other: Infectious titre 2 (H3N2) — Infectious titre 2: 2.5 x 10*4 TCID50/mL
  Arms: Infectious titre 2
Other: Infectious titre 3 (H3N2) — Infectious titre 3: 3.6 x 10*5 TCID50/mL
  Arms: Infectious titre 3
Other: Infectious titre 4 (H3N2) — Infectious titre 4: 4.7 x 10*6 TCID50/mL
  Arms: Infectious titre 4
Other: Infectious titre 5 (H3N2) (Subjects aged 18 to 45 years old) — Infectious titre 5: 3.5 x 10*5 TCID50/mL
  Arms: Infectious titre 5 (age 18 to 45 y)
Other: Infectious titre 5 (H3N2) (Subjects aged 46 to 64 years old) — Infectious titre 5: 3.5 x 10*5 TCID50/mL
  Arms: Infectious titre 5 (age 46 to 64 y)

SUMMARY:
The study will characterise Influenza A/Perth/16/2009(H3N2) virus in healthy participants using the viral challenge model. The study includes two cohorts.

Cohort 1: A randomised, double-blind study of 4 titres of Challenge Virus to determine the optimum titre.

Cohort 2: An open-label extension arm in which all participants will receive the 'optimum' titre as identified from Cohort 1.

DETAILED DESCRIPTION:
Influenza and its associated diseases are a major cause of morbidity and mortality. The United States Advisory Committee on Immunization Practices recommends influenza vaccination for everyone over 6 months of age. The failure of the flu vaccine in 2014-2015 demonstrates the need for a model that allows the rapid development of novel antivirals, universal/intra-seasonal vaccines, immunomodulators, monoclonal antibodies and other novel treatments. Studies using experimental influenza virus infection in human participants have demonstrated that adult volunteers can be infected by nasal inoculation, and experimental infection is safe and not associated with transmission to contacts. The experimental virus is manufactured in compliance with Good Manufacturing Practice for use in the Human Viral Challenge Model.

The investigators chose an H3N2 influenza subtype given that this strain has the most substantial impact in terms of morbidity or mortality annually as described by the Centre for Disease Control . The investigators first subjected the virus batch to rigorous adventitious agent testing, then confirmed the virus to be wild-type by Sanger sequencing and finally determined the virus titres appropriate for human use via the established ferret model. hVIVO team built on its previous experience with other H3N2 and H1N1 viruses to develop this unique model.

The first part of study (Cohort 1) was to determine the safety and optimal virus titre in healthy adult volunteers using our unique clinical quarantine facility in London, UK. After the first part of the study was completed, the study was amended to add an older population group (45-64 years old) in order to characterise the course of infection in an age group better representing the at-risk population.

ELIGIBILITY:
Inclusion Criteria:

* In good health with no history of major medical conditions.
* A total body weight ≥ 50 kg and a BMI of >18.
* Acceptable forms of effective contraception.
* An informed consent document signed and dated by the subject and Investigator.
* Sero-suitable for Challenge Virus.

Exclusion Criteria:

* Subjects who have a significant history of any tobacco use at any time (≥ total 10 pack year history, e.g. one pack a day for 10 years).
* Subjects who have been pregnant within six months prior to the study, or who have a positive pregnancy test at any point in the study.
* Any history or evidence of any clinically significant medical conditions (cardiovascular, gastrointestinal, endocrinological, haematological, hepatic, immunological, metabolic, urological, neurological, psychotic, renal, and/or other major disease or malignancy).
* History or evidence of autoimmune disease or known immunodeficiency of any cause.
* Subjects with any history of asthma, COPD, pulmonary hypertension, reactive airway disease, or chronic lung condition of any aetiology.
* Positive human immunodeficiency virus (HIV), Hepatitis A (HAV), B (HBV), or C (HCV) test.
* Any significant abnormality altering the anatomy of the nose or nasopharynx.
* Any clinically significant history of epistaxis (nose bleeds).
* Any nasal or sinus surgery within six months of inoculation.
* Recurrent history of clinically significant autonomic dysfunction.
* Any abnormal laboratory test or ECG.
* Confirmed positive test for drugs of abuse.
* Venous access deemed inadequate for the phlebotomy and cannulation.
* Any known allergies to the excipients in the Challenge Virus inoculums.
* Health care workers who work in units with severely immuno-compromised patients.
* Evidence of vaccinations within the four weeks prior to Human Viral Challenge or intention to receive travel vaccination before the last study visit.
* Receipt of blood or blood products, or loss (including blood donations) of 450 mL or more of blood, during the 3 months prior to inoculations.
* Presence of significant respiratory symptoms existing on the day of challenge or between admission to the unit and inoculation with virus.
* History suggestive of respiratory infection within 14 days prior to admission to the unit.
* Use within 28 days prior to Human Viral Challenge (Day 0) of nasal steroids * Use within seven days of any other medication or product (prescription or over-the-counter), for symptoms of hay fever, rhinitis, nasal congestion or respiratory tract infection.
* Receipt of systemic: glucocorticoids, antiviral drugs, or immunoglobulins (Igs) or any other cytotoxic or immunosuppressive drug.
* Receipt of any systemic chemotherapy agent at any time.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08-11 (Actual); Study Completion 2014-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Muray, MD, Principal Investigator — Hvivo

REFERENCES:
- [Result] Fullen DJ, Noulin N, Catchpole A, Fathi H, Murray EJ, Mann A, Eze K, Balaratnam G, Borley DW, Gilbert A, Lambkin-Williams R. Correction: Accelerating Influenza Research: Vaccines, Antivirals, Immunomodulators and Monoclonal Antibodies. The Manufacture of a New Wild-Type H3N2 Virus for the Human Viral Challenge Model. PLoS One. 2016 Jun 9;11(6):e0157211. doi: 10.1371/journal.pone.0157211. eCollection 2016. PMID 27280602
- [Derived] Fullen DJ, Noulin N, Catchpole A, Fathi H, Murray EJ, Mann A, Eze K, Balaratnam G, Borley DW, Gilbert A, Lambkin-Williams R. Accelerating Influenza Research: Vaccines, Antivirals, Immunomodulators and Monoclonal Antibodies. The Manufacture of a New Wild-Type H3N2 Virus for the Human Viral Challenge Model. PLoS One. 2016 Jan 13;11(1):e0145902. doi: 10.1371/journal.pone.0145902. eCollection 2016. PMID 26761707

RESULTS

PARTICIPANT FLOW:
Groups:
- Infectious Titre 1: Infectious titre 1:
  6 subjects aged 18 to 45 received 1mL containing 2.8 x 10*3 TCID50
  Infectious titre 1: 2.8 x 10*3 TCID50/mL
- Infectious Titre 2: Infectious titre 2:
  6 subjects aged 18 to 45 received 1mL containing 2.5 x 10*4 TCID50
  Infectious titre 2: 2.5 x 10*4 TCID50/mL
- Infectious Titre 3: Infectious titre 3:
  6 subjects aged 18 to 45 received 1mL containing 3.6 x 10*5 TCID50
  Infectious titre 3: 3.6 x 10*5 TCID50/mL
- Infectious Titre 4: Infectious titre 4:
  6 subjects aged 18 to 45 received 1mL containing 4.7 x 10*6 TCID50
  Infectious titre 4: 4.7 x 10*6 TCID50/mL
- Infectious Titre 5 (18 to 45 Years Old): Infectious titre 5:
  6 subjects aged 18 to 45 received 1mL containing 3.5 x 10*5 TCID50
  Infectious titre 5: 3.5 x 10*5 TCID50/mL
- Infectious Titre 5 (46 to 64 Years Old): Infectious titre 5:
  16 subjects aged 46 to 64 received 1mL containing 3.5 x 10*5 TCID50
  Infectious titre 5: 3.5 x 10*5 TCID50/mL
Period: Overall Study
Arm/Group | Infectious Titre 1 | Infectious Titre 2 | Infectious Titre 3 | Infectious Titre 4 | Infectious Titre 5 (18 to 45 Years Old) | Infectious Titre 5 (46 to 64 Years Old)
Started | 6 | 6 | 6 | 6 | 6 | 16
Completed | 6 | 6 | 6 | 6 | 6 | 16
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Infectious Titre 1: 6 participants aged 18 to 45 inoculated with 1mL containing 2.8 x 10*3 TCID50
- Infectious Titre 2: 6 participants aged 18 to 45 inoculated with 1mL containing 2.5 x 10*4 TCID50
- Infectious Titre 3: 6 participants aged 18 to 45 inoculated with 1mL containing 3.6 x 10*5 TCID50
- Infectious Titre 4: 6 participants aged 18 to 45 inoculated with 1mL containing 4.7 x 10*6 TCID50
- Infectious Titre 5 (18 to 45 Years Old): 6 participants aged 18 to 45 inoculated with 1mL containing 3.5 x 10*5 TCID50
- Infectious Titre 5 (46 to 64 Years Old): 16 participants aged 46 to 64 inoculated with 1mL containing 3.5 x 10*5 TCID50
- Total: Total of all reporting groups
Arm/Group | Infectious Titre 1 | Infectious Titre 2 | Infectious Titre 3 | Infectious Titre 4 | Infectious Titre 5 (18 to 45 Years Old) | Infectious Titre 5 (46 to 64 Years Old) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 16 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 16 | 46
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 3 | 2 | 5 | 17
  Male | 2 | 5 | 4 | 3 | 4 | 11 | 29
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 6 | 6 | 6 | 16 | 46

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Virus Load
Description: Area under the curve (AUC) of the Challenge Viral load, measured by nasopharyngeal swab quantitative polymerase chain reaction [qPCR], from Day 1 to Day 8 post-Viral Challenge. Nasopharyngeal swabs are collected up to 3 times per day ( every 8 hours +/- 30mins)
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: mins*Eq log10 TCID50/mL
Groups:
- Infectious Titre 1: Participants aged 18 to 45 received 1mL containing 2.8 x 10*3 TCID50
- Infectious Titre 2: Participants aged 18 to 45 received 1mL containing 2.5 x 10*4 TCID50
- Infectious Titre 3: Participants aged 18 to 45 received 1mL containing 3.6 x 10*5 TCID50
- Infectious Titre 4: Participants aged 18 to 45 received 1mL containing 4.7 x 10*6 TCID50
- Infectious Titre 5 (18 to 45 Years Old): Participants aged 18 to 45 received 1mL containing 3.5 x 10*5 TCID50
- Infectious Titre 5 (46 to 64 Years Old): Participants aged 46 to 64 received 1mL containing 3.5 x 10*5 TCID50
Arm/Group | Infectious Titre 1 | Infectious Titre 2 | Infectious Titre 3 | Infectious Titre 4 | Infectious Titre 5 (18 to 45 Years Old) | Infectious Titre 5 (46 to 64 Years Old)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 16
mins*Eq log10 TCID50/mL | -2081.98 (869.61) | 18,973.90 (1048.23) | 15,944.09 (13751.39) | 12,201.14 (8877.43) | 9563.26 (10,536.96) | 11,710.28 (11833.87)

2. Other Pre Specified Outcome: Incidence (Number and Percentage [%]) of Viral Challenge Emergent Adverse Events
Time Frame: 8 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events are collected throughout the study from screening to last study visit (108 days)
Groups:
- Infectious Titre 1: Infectious titre 1:
  6 participants aged 18 to 45 were inoculated with 1mL containing 2.8 x 10*3 TCID50
  Infectious titre 1: 2.8 x 10*3 TCID50/mL
- Infectious Titre 2: Infectious titre 2:
  6 participants aged 18 to 45 were inoculated with 1mL containing 2.5 x 10*4 TCID50
  Infectious titre 2: 2.5 x 10*4 TCID50/mL
- Infectious Titre 3: Infectious titre 3:
  6 participants aged 18 to 45 were inoculated with 1mL containing 3.6 x 10*5 TCID50
  Infectious titre 3: 3.6 x 10*5 TCID50/mL
- Infectious Titre 4: Infectious titre 4:
  6 participants aged 18 to 45 were inoculated with 1mL containing 4.7 x 10*6 TCID50
  Infectious titre 4: 4.7 x 10*6 TCID50/mL
- Infectious Titre 5 (Aged 18 to 45): 6 participants aged 18 to 45 were inoculated with 1mL containing 3.5 x 10*5 TCID50
  Infectious titre 5: 3.5 x 10*5 TCID50/mL
- Infectious Titre 5 (Aged 45 to 64): 16 participants aged 46 to 64 were inoculated with 1mL containing 3.5 x 10*5 TCID50
  Infectious titre 5: 3.5 x 10*5 TCID50/mL
Arm/Group | Infectious Titre 1 | Infectious Titre 2 | Infectious Titre 3 | Infectious Titre 4 | Infectious Titre 5 (Aged 18 to 45) | Infectious Titre 5 (Aged 45 to 64)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/16
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6 | 3/6 | 2/6 | 2/6 | 10/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infectious Titre 1 (N=6) | Infectious Titre 2 (N=6) | Infectious Titre 3 (N=6) | Infectious Titre 4 (N=6) | Infectious Titre 5 (Aged 18 to 45) (N=6) | Infectious Titre 5 (Aged 45 to 64) (N=16)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Spirometry abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALT increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AST increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vital capacity decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes